CLINICAL TRIAL: NCT07067411
Title: The Effect of an Education Program Given to Patients With Gestational Diabetes Mellitus Using a Gamification Technique on Diabetes Self-Management
Brief Title: Gamified Education for Diabetes Self-Management in GDM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Begum Kirik, Lecturer, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YU-HEM-BK-01
Record Dates: First submitted 2025-07-02; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: gestational diabetes; self-management; gamification; nursing
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: The participants in the intervention group will be shared with an information video link created by the researcher, no longer than five minutes, one day before each game. The participants in the intervention group will be given the game link after watching the information video. The order of the five games planned to be included in the research is; "What is Gestational Diabetes?", "Nutrition Education", "Complication Precautions", "Medical Treatment Applications" and "Physical Activity".
Who Masked: Investigator
Masking Description: After the pre-test application, participants will be assigned equally to the experimental and control groups. Participants to be included in the study will be assigned to the experimental and control groups by block randomization using a computer-aided randomization application (www.randomizer.org) and will be numbered. In addition, the group matching method will be used in the study to ensure homogeneity in the experimental and control groups. With this method, the groups will be arranged to be similar in terms of factors such as age, gestational week, and educational status, so that comparisons between the two groups will be made only on the effects resulting from the independent variable. This approach will increase the validity of the study and the reliability of the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The group participating in the Education Program Given with Gamification Technique (Experimental): 39 participants were assigned as a result of randomization. Participants receiving care through games.
  Interventions: Behavioral: Education Program Using Gamification on GDM
- Control (No Intervention): 39 participants were assigned as a result of randomization. Receiving only routine care.

INTERVENTIONS:
Behavioral: Education Program Using Gamification on GDM — The five games planned to be used in the study are; "What is Gestational Diabetes?", "Nutrition Education", "Complication Precautions", "Medical Treatment Applications" and "Physical Activity". The creation and implementation of these games will be done through the "Genially" platform. The Genially platform is an easy-to-use and free web tool used to create interactive visual content. The platform includes features such as sharing or downloading via website, social media or e-mail by adding animations, effects, sounds and interactive elements. In addition, the performances of the people who share the created content can be tracked and feedback can be obtained. At the beginning of the games planned to be used in the study, an informative video of not more than five minutes on the subject created by the researcher will be shared. National and international guidelines will be taken into consideration in the creation of these videos. One day after the informative video is
  Arms: The group participating in the Education Program Given with Gamification Technique

SUMMARY:
Gestational diabetes mellitus (GDM) is a serious public health problem characterized by hyperglycemia that develops during pregnancy and causes significant short- and long-term health risks for both the mother and the fetus. Lifestyle changes, especially appropriate diet and exercise practices and glycemic control are among the basic approaches in GDM management. However, the individual's adoption and sustainability of these approaches are often insufficient, and the individual's participation in treatment and motivation levels may be limited.

When the literature is examined, it has been proven that gamification-based interventions, especially in individuals with type 2 diabetes, have positive effects such as increasing the level of knowledge, encouraging physical activity and improving glycemic control. However, the lack of gamification-based nursing interventions specific to women with GDM is striking. The fact that there is no standardized nursing protocol specific to GDM management in our country makes the literature gap in this area even more evident.

This study aims to develop health behaviors in individuals with GDM through a gamified training program to be developed based on the Information-Motivation-Behavioral Skills (IMB) model. Thanks to the innovative structure of gamification, it is aimed not only to increase the knowledge level of individuals, but also to increase their motivation and make behavioral changes permanent. Thus, the active participation of the individual in the treatment process will be encouraged and the self- management skills will be strengthened.

This research will be an important step in terms of the integration of digitalization and patient-centered approaches in nursing practices, as well as indirectly contributing to the protection and development of public health. While the training program has the potential to increase the quality of life at the individual level, it will also allow the development of an original and structured nursing care intervention that can be used in GDM management.

This study aims to fill an important gap in the literature, to disseminate innovative practices in the field of nursing, and to support healthy pregnancy outcomes at the social level. For this reason, the purpose of the research was planned to examine the effect of the training program applied to women with gestational diabetes with the gamification technique based on the information-motivation-behavior (IMB) model on diabetes self-management.

ELIGIBILITY:
Inclusion Criteria:

* Those who speak Turkish,
* Literate,
* Between the ages of 18 and 40,
* Those diagnosed with Gestational Diabetes Mellitus (based on a single-stage and/or two-stage oral glucose tolerance test between the 24th and 28th weeks),
* Those with a singleton pregnancy,
* Pregnant women who have not been previously diagnosed with diabetes,
* Those who do not have a chronic disease diagnosed by a doctor (hypertension, cardiovascular diseases, kidney diseases, anemia, thyroid and autoimmune diseases),
* Those who do not have any other pregnancy-related problems (gestational hypertension, preeclampsia, gestational thyroiditis, etc.),
* Those who do not have a physical disability,
* Pregnant women who have access to the internet via phone or computer will be included in the sample.

Exclusion Criteria:

* Those who cannot read or write,
* Those with threatened premature labor (PTD), premature membrane rupture (PROM), preeclampsia; risky pregnancy conditions,
* Intrauterine mortal fetus,
* Those who have experienced significant losses in the last 3 months (divorce, death of a loved one, etc.),
* Those with moderate to severe (over 14 points) depressive symptoms as a result of the Patient Health Questionnaire-8 (PHQ-8) will be considered as a risk group and will not be included in the sample.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Self-Efficacy Scale in Gestational Diabetes | through study completion, an average of 1 year
  The validity and reliability of the "Self-Efficacy Scale in Gestational Diabetes" was determined by Polat and Ünsal Avdal and it was concluded that it is a valid and reliable measurement tool. The Self-Efficacy Scale in Gestational Diabetes (SESGD) is a five-point Likert-type scale consisting of four sub-dimensions. The sub-dimensions of the scale are; ''Diet-Weight Management'', ''Complication Precautions'', ''Adherence to Nutrition Education'' and ''Medical Treatment Applications''. The total Cronbach alpha value of the scale was determined as 0.654. The scale includes positive and negative statements. Reverse and forward coding is done during the analysis. It can be thought that as the score to be obtained from the scale increases as a result of the coding of positive and negative statements in the scale, the individual's self-efficacy will increase and that he/she will be able to effectively take care of himself/herself as a result of the education he/she receives.

OTHER OUTCOMES:
International Physical Activity Questionnaire Short Form-Turkish version (IPAQ) | through study completion, an average of 1 year
  For the analysis of IPAQ data, it is evaluated as "walking: 3.3 MET", "moderate physical activity: 4.0 MET", "vigorous physical activity: 8.0 MET". Daily and weekly physical activity levels are calculated using these values. As the MET value increases, the physical activity level increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Women and Children Diseases Traning and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No